CLINICAL TRIAL: NCT07006805
Title: RESET-MS: A Phase 1/2, Open-Label Study to Evaluate the Safety and Efficacy of Autologous CD19-specific Chimeric Antigen Receptor T Cells (CABA-201) in Participants With Multiple Sclerosis
Brief Title: RESET-MS: A Study to Evaluate the Safety and Efficacy of CABA-201 in Participants With Multiple Sclerosis
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cabaletta Bio (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CAB-201-005
Record Dates: First submitted 2025-04-22; First posted 2025-06-05 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Relapsing Multiple Sclerosis (RMS); Progressive Multiple Sclerosis (PMS); Multiple Sclerosis - Relapsing Remitting; Multiple Sclerosis; Multiple Sclerosis (Relapsing Remitting); Multiple Sclerosis (MS) - Relapsing-remitting; Progressive Multiple Sclerosis
Keywords: CABA-201; Rese-cel; autoimmune disease; anti-CD19 CAR-T therapy; cellular therapy; Multiple Sclerosis; Relapsing MS; RRMS; Progressive MS; PPMS; SPMS; Neurology; Resecabtagene autoleucel
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive; Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis; Autoimmune Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Relapsing MS Cohort (Experimental)
  Interventions: Biological: CABA-201
- Progressive MS Cohort (Experimental)
  Interventions: Biological: CABA-201

INTERVENTIONS:
Biological: CABA-201 — Single intravenous infusion of CABA-201 following preconditioning with fludarabine and cyclophosphamide

SUMMARY:
RESET-MS: A Phase 1/2 Open-Label Study to Evaluate the Safety and Efficacy of Autologous CD19-specific Chimeric Antigen Receptor T cells (CABA-201) in Participants with Multiple Sclerosis

DETAILED DESCRIPTION:
This is a Phase 1/2, open-label study designed to evaluate the safety, tolerability, and efficacy of different doses of CABA-201 in adult participants with MS to determine an appropriate dose for future studies. Any participant who receives CABA-201 will be followed after infusion for 156 weeks. Two cohorts of participants will be studied based upon their MS diagnosis.

* Relapsing MS Cohort (RMS Cohort): Participants with active relapsing MS, including relapsing remitting MS (RRMS) and relapsing secondary progressive MS (SPMS) that is treatment-resistant
* Progressive MS Cohort (PMS Cohort): Participants with worsening progressive MS, including primary progressive MS (PPMS) or non-relapsing SPMS that is treatment-resistant

The study will consist of 2 parts: Part A (dose escalation) and Part B (dose expansion).

ELIGIBILITY:
Inclusion Criteria

The main inclusion criteria include the following:

* Able to provide informed consent.
* Age ≥18 and ≤60 years of age.
* Diagnosis of MS per the revised 2017 McDonald criteria (Thompson et al, 2018).
* For participants with relapsing forms of MS only (RMS Cohort):

  1. Moderate degree of previously accumulated disability as measured by the Expanded Disability Status Scale (EDSS)
  2. Documentation of clinical relapse or a positive historical gadolinium (Gd)-enhancing magnetic resonance imaging (MRI) scan prior to Screening
  3. Prior treatment with a high-efficacy therapy or prior treatment failure of oral therapies
* For participants with progressive forms of MS only (PMS cohort):

  1. Moderate Disability as measured by EDSS
  2. Presence of abnormal function on protocol specified EDSS Functional Systems Scale
  3. Objective worsening of disease prior to Screening while on standard of care therapy
* Clinical stability by vital signs assessment at the time of screening

Exclusion Criteria

The main exclusion criteria include the following:

* History of fulminant MS
* Clinically significant concomitant central nervous system pathologies which, in the Investigator's judgement, may confound the ability to interpret study results or complicate identification or evaluation of neurotoxicity, including but not limited to:

  1. Any history of seizure disorder, even if well-controlled on antiepileptics
  2. History of progressive multifocal leukoencephalopathy
* Active, inflammatory autoimmune disorder other than MS requiring immunomodulatory therapies

  a. Positive human immunodeficiency virus (HIV), hepatitis C virus (HCV) antibody, or hepatitis B surface antigen test, or evidence of active or chronic tuberculosis (TB) at Screening or other chronic viral infections as described in the protocol
* Use of the following therapies:

  1. Any prior or concurrent exposure to mitoxantrone, alemtuzumab, total lymphoid irradiation
  2. Cladribine within 1 year of Screening
  3. Any investigational agent within 4 weeks or 5 half-lives of Screening, whichever is longer
  4. Other pre-specified Disease-Modifying Therapies be discontinued by the time of pre-conditioning or earlier as described in the protocol
* Known malignancy or a history of malignancy
* Current symptoms of severe, progressive, or uncontrolled renal, hepatic, hematological, gastrointestinal, pulmonary, psychiatric, cardiac, or concomitant neurological disease, including severe (requiring medical intervention) and uncontrolled infections
* Chronic pulmonary disease
* Impaired cardiac function or clinically significant cardiac disease
* Prior engineered T cell therapy involving permanent gene modification
* Prior solid organ (heart, liver, kidney, lung) transplant or hematopoietic stem cell transplant.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Primary (Part A: Dose Escalation) incidence and severity of adverse events | Up to 28 days after CABA-201 infusion
  An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal result of an investigation), symptom, or disease (new or exacerbated) temporally associated with the use of study treatment. The term AE is used to include both serious and non-serious AEs.
Primary (Part B: Dose Expansion) incidence of and severity of adverse events in order to confirm the dose(s) of CABA-201 | Up to 28 days after CABA-201 infusion
  An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal result of an investigation), symptom, or disease (new or exacerbated) temporally associated with the use of study treatment. The term AE is used to include both serious and non-serious AEs.

SECONDARY OUTCOMES:
Part A and Part B: To evaluate the incidence and severity of adverse events | Up to 156 weeks after CABA-201 infusion
  An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal result of an investigation), symptom, or disease (new or exacerbated) temporally associated with the use of study treatment. The term AE is used to include both serious and non-serious AEs.
Part A and Part B: To characterize the pharmacodynamics (PD) | Up to 156 weeks after CABA-201 infusion
  Levels of B cells in the blood
Part A and Part B: To characterize the pharmacokinetics (PK) | Up to 156 weeks after CABA-201 infusion
  Levels of CABA-201-positive T cells in the blood
Part A and Part B: To evaluate disease related biomarkers | Up to 156 weeks after CABA-201 infusion
  Levels of MS biomarkers in the blood and CSF
Part A and Part B: To evaluate the effects of CABA-201 on MS disease activity as measured by Magnetic Resonance Imaging (MRI) | Up to 156 weeks after CABA-201 infusion
  Incidence of accumulated MS-related lesions
Part A and Part B: The effects of CABA-201 on MS disease activity as measured by EDSS | Up to 156 weeks after CABA-201 infusion
  The EDSS is a scale for assessing neurologic impairment in MS. Values are from 0 points (normal neurological examination) up to 10 points (death). Higher scores represent increased disability.
Part A and Part B: To evaluate the effect of CABA-201 on use of subsequent MS-related therapy | Up to 156 weeks after CABA-201 infusion
  Proportion of participants who require no subsequent MS-related immunomodulatory therapy
Part A and Part B: To evaluate the effect of CABA-201 on patient reported and health outcomes as measured by SF-36 v2 | Up to 156 weeks after CABA-201 infusion
  Change in SF-36 v2

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Chair — Cabaletta Bio

IPD SHARING:
Plan to Share IPD: No